CLINICAL TRIAL: NCT05798299
Title: Exploratory Randomized Controlled Trial of a Child-centered Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children (UP-C/C)
Brief Title: Efficacy Study of a Child-centered Version of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Children
Acronym: UP-C/C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lisbon (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); University of Coimbra (Other)
Responsible Party: Principal Investigator, Ana Isabel de Freitas Pereira, Principal Investigator, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.06835.BD
Record Dates: First submitted 2023-03-17; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Emotional Disorders; Childhood Anxiety; Childhood Depression
Keywords: Randomized controlled trial; Anxiety Disorders; Mood disorders; Transdiagnostic Intervention; UP-C; UP-C/C; Parenting
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP-C/C (Experimental): UP-C/C intervention - 15 weekly sessions for children; 3 group sessions for parents; 1 family meeting before exposure sessions.
  Interventions: Behavioral: Arm 1: Transdiagnostic intervention
- Coping Cat, Group Format (Active Comparator): Coping Cat in group format intervention - 16 weekly sessions for children; 2 individual sessions for parents.
  Interventions: Behavioral: Arm 2: Anxiety-focused intervention

INTERVENTIONS:
Behavioral: Arm 1: Transdiagnostic intervention — The UP-C/C consists of 15 weekly sessions for children, each lasting 90 minutes. It is also composed by three sessions for parents and a meeting with the family prior to the exposure sessions. Parents have access to weekly psychoeducational material (in written and in video format) and help the children with homework completion.
  Other Names: UP-C/C; Unified Protocol for Children - Child-Centered Version; Emotion Detectives - Child-Centered Version
  Arms: UP-C/C
Behavioral: Arm 2: Anxiety-focused intervention — The Coping Cat in group format is a cognitive-behavioral evidence-based intervention for anxiety problems. It is composed by 16 90-minute sessions for children and two parenting sessions.
  Arms: Coping Cat, Group Format

SUMMARY:
The UP-C is a manualized, cognitive-behavioral, and emotion-focused group intervention with a transdiagnostic approach aimed at the treatment of emotional problems (i.e., anxiety and depression) in children aged 7 to 12 years old. This psychological intervention mainly focuses on reducing the intensity and frequency of strong and aversive emotional experiences in children through the development of skills that allow them to face these emotions in a more adaptive way.

By targeting the factors common to emotional disorders (avoidance, emotional reactivity, affective intolerance) we believe this intervention might increase the effectiveness of the treatment of these difficulties (mainly in the cases where comorbidity is present). It may also contribute to therapists' expertise when dealing with different emotional disorders, by not requiring the simultaneous mastery of multiple interventions, to a reduction of costs associated with training and to the planning of more individualized and flexible interventions. This approach could help to make interventions suitable for a set of problems more accessible to the public - which is particularly relevant to the Portuguese context. Thus, to better adapt to the limitations existent in mental health services in Portugal, a modified version of the UP-C was developed by reducing the number of sessions for parents.

The current study seeks to understand whether this adapted version of the UP-C - the UP-C/C - less demanding in terms of resources required for its application, is effective in reducing children's emotional symptomatology and produces changes on maladaptive parenting strategies used by parents. This version is mostly centered on the child, who participates in 15, 90 minutes, group sessions. In this version of the program, the parents adopt the role of "cotherapists", and support homework completion at home by the child. They also have access to psychoeducational material (in video and written format). Additionally, the UP-C/C includes three parental sessions that focus on parenting strategies shown to be useful in challenging situations. This study also seeks to evaluate child and parent involvement in the intervention and understand its predictors.

These are the specific objectives of the study:

1. To evaluate the efficacy of the UP-C/C through a Randomized Controlled Clinical Trial with two conditions (UP-C/C and Coping Cat in group format) on the primary outcomes (child's anxiety and depression symptoms, interference of anxiety and depression in the child's school, social and family functioning), secondary (quality of life, emotional expression and cognitive errors), and on the transdiagnostic factors (avoidance, emotional reactivity, affective intolerance) and on the parental variables (parents' emotional behaviors, orientation towards the child's emotions, symptoms of anxiety and depression);
2. To evaluate the involvement of the child and parents in the program (attendance, dropout, active participation) and find out its predictors (age; intensity of symptoms; readiness for change; therapeutic alliance; expectations regarding the intervention).

The main hypothesis of the study, relating to the efficacy study, is the following:

- UP-C/C is expected to have equivalent results to Group Coping Cat in outcomes related to anxiety and quality of life and superior results in outcomes related to depression and transdiagnostic mechanisms.

DETAILED DESCRIPTION:
Participants will be recruited from schools located in Lisbon's metropolitan area (Portugal). The selection of participants will be carried out through a two-phase screening, after parental consent and assent from the children are obtained. In both phases, the children will complete a questionnaire that assesses symptoms of anxiety and depression. Children whose score in the screening of anxiety symptoms is in a percentile equal to or greater than 80 will be selected at both assessment times. Families of children selected through the screening are invited to an individual assessment session. In this session, a brief set of questions to parents is asked to ensure their child's eligibility, and current difficulties are explored in more detail. If the necessary criteria are met, the pre-intervention evaluation processes take place (child and caregivers complete a set of measures).

To access the efficacy of the UP-C/C, this intervention will be compared with a cognitive-behavioral intervention previously shown to be effective in the treatment of anxiety disorders, the Coping Cat program in a group format. Thus, once the recruitment and evaluation of eligibility criteria is finished, the children and their parents will be randomly allocated to one of two conditions:

1. experimental group (i.e., children and parents who benefit from the UP-C/C program);
2. control group (i.e., children who benefit from the Coping Cat, group format).

In both conditions, 15/16 weekly sessions with the children will take place in groups of 5 to 7 participants. Therapist's and children's manuals are available. The groups will be conducted by clinical psychologists integrated in the research team. All therapists received training to conduct the intervention and will receive weekly supervision by the project supervisor. Every session will be observed and evaluated by an external observer through a checklist.

Regarding the primary and secondary outcomes, transdiagnostic mechanisms and parental variables, the study includes 5 assessment times - at pre-intervention, 6 weeks after the start of the intervention, after the intervention ends and at two follow-ups, 3 and 6 months after the end of the intervention. The variables related to the therapeutic process are evaluated at each session (active participation, assessment of program conduction, therapeutic alliance) and in the 1st session (readiness for change). Informed consent, from the parents and the children, will be sought at each assessment time. Consent protocol includes a paragraph, that explains how data will be recorded and who has access to it. Only information relevant to the study is collected.

For the analysis of the effects of the intervention, a multivariate analysis of variance (MANOVA) (SPSS 26.0) will be used. To assess participants' engagement in the UP-C/C, data will be collected from all sessions and percentages of attendance and dropout will be calculated. ANOVA analysis of variance and Chi-Square tests (SPSS 26.0) will be used to examine differences between the Experimental Group and the Control Group in attendance/active participation and dropout, respectively. To explore predictors of attendance/active participation and dropout Multiple Regressions and Logistic Regressions (SPSS 26.0) will be used, respectively.

Assuming a mean effect size of 0.4 on improvement in depressive symptomatology, an alpha=0.05, and power=0.8, for a 2-group design with 5 repeated measures, the total sample size required is 80 (G*Power). Given an expected dropout of 17%, it will be necessary to recruit a minimum of approximately 94 children. Thus, a sample of 47 children in the experimental group and 47 in the control group is expected. 7 UP-C/C groups with a maximum number of 7 children will be conducted. To allow for a satisfactory number of participants, the therapeutic groups will be carried out in two periods (March 2023 to July 2023 and October 2024 to February 2024).

Missing data due to participant's dropout will be handled by intention-to-treat principles, estimated using the last observation carried forward (LOCF) method.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12;
* Children whose score in the screening of anxiety symptoms is in a percentile equal to or greater than 80;
* Speaking, reading and understanding Portuguese;

Exclusion Criteria:

* Diagnosis of a psychotic disorder, bipolar disorder, intellectual disability or autism spectrum disorder;
* Severe current suicidal/homicidal ideation;
* The child is being subjected to a not yet stable dose of a psychotropic or other type of medication (i.e., modified less than 1 month prior to baseline assessment);
* The child or parents are not fluent in the Portuguese language;
* The child is benefiting from another psychological intervention;
* Presence of the parents and the child cannot be guaranteed in most of the intervention and assessment sessions; the presence of the parents is only required in the parenting sessions and in the evaluation sessions (week 6, after the intervention, and two follow-ups).

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the children's anxiety and depression | Recruitment/Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured with the Revised Children's Anxiety and Depression Scale (RCADS) (Child and Parent Version)
  Child version: Self-report questionnaire composed by 47 items and 6 subscales, including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive-compulsive disorder, and major depression. It also includes a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales).
  Parent version: Measure completed by the parents that includes 6 subscales to assess the child's anxiety and depression symptoms.
Changes in the children's severity of psychopathology and improvement | Baseline, Mid-treatment (6 weeks); Post treatment (15 weeks)
  Measured with an adaptation of the Clinical Global Impression (CGI). Brief assessment of the patient's global functioning before and after the intervention, the CGI is composed by an illness' severity scale and a scale evaluating changes in the patient's symptoms relative to their condition at the start of the intervention. Higher scores are indicative of higher severity of psychopathology.
Changes in the child's anxiety life interference | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured with the Child Anxiety Life Interference Scale (Child and Parent Versions)
  Child version: Questionnaire for evaluating the influence of the child's symptoms on their school, social and family functioning.
  Parent version: Measure for assessing the influence of the child's symptoms on their school, social and family functioning through parental report.

SECONDARY OUTCOMES:
Changes in the children's behavioral avoidance | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured with the Child- and Parent-Report Measures of Behavioral Avoidance Related to Childhood Anxiety Disorders (CAMS and CAMP). Higher scores indicate higher levels of children's behavioral avoidance.
Changes in the children's negative affect | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured with the Positive and Negative Affect for Children (PANAS-C). PANAS-C is composed by 10 items for the assessment of Positive Affect and Negative Affect, organized in two scales. Higher scores are indicative of higher levels of children's positive and negative affect, respectively.
Changes in the children's anxiety sensitivity | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by Children's Anxiety Sensitivity Inventory-Revised (CASI-R). Higher scores are indicative of higher levels of anxiety sensitivity.
Changes in the children's cognitive distortions | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by the Children's Negative Cognitive Error Questionnaire (CNCEQ). The CNCEQ assesses four types of cognitive errors and yields a Total Score for each type of cognitive error, a Total Score for areas of content and a Total Score for cognitive errors. Higher values are indicative of a greater presence of cognitive errors.
Changes in the children's emotional expression and emotion awareness | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by the Emotional Expression Scale for Children (EESC). In this measure, higher scores correspond to higher levels of difficulties in children's emotional expression and emotion awareness.
Changes in the children's life quality | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by the Kidscreen-10 index (parent version), a brief measure that assesses the quality of life of the children through parental report.
Changes in parent's anxiety | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks); Follow-up (3 and 6 months)
  Measured by the Generalized Anxiety Disorder Scale (GAD-7), a brief self-report questionnaire with 7 items that assesses the presence of anxiety symptoms. Higher scores are indicative of higher levels of anxiety.
Changes in parent's depression | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks); Follow-up (3 and 6 months)
  Measured by the Patient Health Questionnaire 9 (PHQ-9) that evaluates symptoms of major depression through 9 items. Higher scores are indicative of higher levels of depression.
Changes in parental overprotection | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 months and 6 months)
  Measured by the Parental anxiety and overprotection scale (PAOS). Higher scores are indicative of higher levels parental overprotection.
Changes in parental inconsistency and permissiveness | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by Parenting Styles & Dimensions Questionnaire. Only the permissiveness subscale will be used. Higher scores are indicative of higher levels of parental inconsistency and permissiveness.
Changes in parental criticism | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by the EMBU-P, a questionnaire that assesses parental styles. In the current study, only the rejection subscale will be used, which assesses parental rejection and criticism. Higher scores indicate higher levels of rejection and parental criticism.
Changes in the modeling of negative emotions | Baseline, Mid-treatment (6 weeks), Post-treatment (15 weeks), Follow-up (3 and 6 months)
  Measured by The Parent Emotion Regulation Scale (PERS). In the present study only parents' lack of emotional control scale will be used, which assesses the lack of ability of parents to modulate their own negative emotions in the presence of the child. Higher scores are indicative of higher levels of modeling of negative emotions.

OTHER OUTCOMES:
Changes in the Principal Problems | Baseline; during the intervention (up to 16 weeks); post-intervention
  Measured with the weekly child and parent assessment form of the child's main problems, identified by the parents and children in the pre-treatment evaluation session.
Parent's and children's evaluation of program materials | During the intervention (up to 16 weeks)
  Measured with a feedback form for parents regarding the materials/session - learning and its importance, strategies considered useful, ability to support the child with homework, accomplishment of tasks, difficulties experienced,
  Measured with a feedback form for children regarding the session - enjoyment, learning and its importance, strategies considered useful.
Motivation to change scale - parents and children | Baseline; mid-intervention before exposure sessions
  Measured with a brief 6-item form, the Motivation for Change Rating Scale, for children and parents, that assesses motivation for change.
Children's involvement evaluation | During the intervention (up to 16 weeks)
  Measured with a form that assesses the child's involvement in in-session and out-of-session activities, and their mastery of the skills learned, and the children's rapport with the therapist and other children, by the therapist.
Weekly program assessment | During the intervention (up to 16 weeks)
  Measured with a weekly evaluation form of the attendance of the participants, fulfillment of the goals defined for each activity and of the dynamization by the therapist.
Parent's and Children's Involvement in Therapy | During the intervention (up to 16 weeks)
  Measured with The Parent's and Children's Involvement in Therapy Scale (PIRS and CIRS, respectively) - measures composed of 10 items that assess the involvement of the child and parents in the intervention session. They are composed of items related to active involvement (behaviors that demonstrate the child's active participation in tasks) and items related to negative involvement (behaviors that demonstrate avoidance or withdrawal from the session's tasks).
Therapeutic Alliance | During the intervention (up to 16 weeks)
  Measured with the Therapy Process Observation Coding System-Alliance Scale, a 9-item instrument that provides an objective description of the therapeutic alliance between child and clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Psychology, University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No